CLINICAL TRIAL: NCT01640756
Title: A Prospective, Multicenter Clinical Trial Designed to Evaluate the Safety and Performance of the AqueSys Microfistula Implant in Subjects With Refractory Glaucoma
Brief Title: AqueSys Microfistula Implant in Refractory Glaucoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AqueSys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P11-001
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Glaucoma; Glaucoma, Open-Angle
Keywords: Glaucoma Implant; Trabeculectomy; POAG
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AqueSys Microfistula Implant (Experimental)
  Interventions: Device: AqueSys Microfistula Implant

INTERVENTIONS:
Device: AqueSys Microfistula Implant — Placement of the AqueSys Microfistula Implant in the study eye

SUMMARY:
To establish the safety and performance of the AqueSys Microfistula Implant in eyes with refractory glaucoma.

DETAILED DESCRIPTION:
A prospective, multi-center, single arm, open-label clinical trial to evaluate the safety and IOP lowering performance of the AqueSys Microfistula Implant in refractory glaucoma patients who have previously failed a glaucoma procedure and who are not well-controlled on IOP lowering medications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Refractory Glaucoma
* Maximally-tolerated medicated IOP at two preoperative visits of ≥20 mmHg and ≤35 mmHg
* Visual field mean deviation score of -3 dB or worse
* Shaffer Angle Grade ≥ 3
* Area of free, healthy and mobile conjunctiva in the targeted quadrant

Exclusion Criteria:

* Active Neovascular Glaucoma
* Previous glaucoma shunt/valve in the targeted quadrant
* History of corneal surgery, opacities or disease/pathology
* Anticipated need for ocular surgery
* Non-study eye with BCVA of 20/200 or worse

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a 20% or greater reduction in IOP from baseline on the same or less number of medications | 12 Months

SECONDARY OUTCOMES:
Mean change in IOP from baseline | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Lewis, M.D., Study Chair — Grutzmacher and Lewis Surgical Eye Specialists
Locations (14):
- United States (14):
  - Vold Vision, PLLC, Fayetteville, Arkansas
  - USC Eye Institute, University of Southern California, Los Angeles, California
  - Scripps Clinic, San Diego, California
  - Ophthalmic Consultants of Connecticut, Fairfield, Connecticut
  - Bascom Palmer Eye Institute, University of Miami, Miami, Florida
  - Stiles Eyecare Excellence and Glaucoma Institute, Overland Park, Kansas
  - Minnesota Eye Consultants, PA, Bloomington, Minnesota
  - Eye Care Associates & Glaucoma Consultants of Long Island, Bethpage, New York
  - New York Eye and Ear Infirmary, New York, New York
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Texan Eye, Austin, Texas
  - Glaucoma Associates of Texas, Dallas, Texas
  - UVA Eye Clinic, University of Virginia, Charlottesville, Virginia
  - Spokane Eye Clinic, Spokane, Washington